CLINICAL TRIAL: NCT03453528
Title: Investigation of PSMA PET/CT as an Imaging Biomarker in Solid Tumors
Acronym: BASKET PSMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRST100.34
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Prostate-specific Membrane Antigen; mCRPC or Advanced/Metastatic Solid Tumors
Keywords: mCRPC or advanced/metastatic solid tumors; Prostate-specific membrane antigen
MeSH Terms: interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA (Experimental): 68Ga-PSMA
  Interventions: Drug: 68Ga-PSMA

INTERVENTIONS:
Drug: 68Ga-PSMA — 68Ga-PSMA will be injected intravenously via an indwelling catheter in an antecubital vein; (68Ga-PSMA activity: min 100 MBq - max 200 MBq, weighted activity: 2.0 MBq/Kg).

SUMMARY:
multi-centre, prospective, diagnostic trial to evaluate the Prostate-Specific Membrane Antigen (PSMA-antigen) over-expression in metastatic castration resistant prostate cancer (mCRPC) and in advanced/metastatic solid tumors patients.

DETAILED DESCRIPTION:
Multi-centre, prospective, diagnostic trial to evaluate the Prostate-Specific Membrane Antigen (PSMA-antigen) over-expression in metastatic castration resistant prostate cancer (mCRPC) and in advanced/metastatic solid tumors patients.

The primary objective of this study is to evaluate the detection rate of PSMA PET/CT, defined as the ratio of PSMA-positive patients and the total number of cancer patients with known advanced/metastatic disease that performed a PSMA PET/CT as part of the present study. A positive patient is defined as a patient with at least one PSMA-positive lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mCRPC or advanced/metastatic solid tumors;
2. Male or Female, aged >18 years;
3. Written informed consent;
4. Relapse or progression of disease on CT scan and / or MRI;
5. If female of childbearing potential, highly effective birth control methods according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials" (2014_09_15 section 4.1) are mandatory, beginning at the screening visit and continuing until 6 months following last 68Ga-PSMA PET/CT.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

1. Pregnancy / Nursing;
2. Participation in another clinical trial with any investigational agents within 30 days prior to study entry
3. Medical or psychological conditions that would not allow the participant to understand, or sign the informed consent.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to 68Ga-PSMA or other agents used in the study.
5. inability to remain still for the entire duration of the exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1225 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
detection rate of 68Ga-PSMA PET/CT | up to 36 months
  the proportion of 68Ga-PSMA- positive patients and the total number of recruited patients in two groups population's (metastatic castration-resistance prostate cancer and various origin solid tumors).

SECONDARY OUTCOMES:
Safety is defined as the number and percentage of treated patients undergoing grade 1 to 4 adverse events according to CTCAE version 4.03 | up to 36 months
  Safety is defined as the number and percentage of treated patients undergoing grade 1 to 4 adverse events according to CTCAE version 4.03
Lesion detection rate stratified per tumor histotypes | up to 36 months
  Proportion of positive patients on total number who underwent 68Ga-PSMA PET/CT stratified for tumor histotypes;
Lesion detection rate stratified for different lesion sites | up to 36 months
  Proportion of positive patients on total number who underwent 68Ga-PSMA PET/CT stratified for different lesion sites;
Changes in 68Ga-PSMA uptake in patients with other solid tumors who receive anti-angiogenetic therapies according to objective clinical response; | up to 36 months
  Changes in 68Ga-PSMA uptake in patients and correlation with clinical response to 177Lu-PSMA therapy for prostate cancer, or other angiogenic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Caroli, MD, Study Chair — IRST IRCCS
Locations (1):
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC, Italy